CLINICAL TRIAL: NCT04109287
Title: Haemodynamic Changes in Femoral-popliteal Bypass Grafts With the Use of Neuromuscular Electrical Stimulation.
Brief Title: Blood Flow Changes in Femoral-popliteal Bypass Grafts After Neuromuscular Electrical Stimulation (NMES).
Acronym: HAEMUS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19CX5468
Record Dates: First submitted 2019-09-23; First posted 2019-09-30 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Peripheral Arterial Disease; Peripheral Artery Disease; Peripheral Vascular Disease; Femoral Popliteal Occlusion
Keywords: Femoral-popliteal; Bypass; Graft; PAD; PVD; NMES; Time-averaged mean velocity; Volume flow rate; Volume flow; TAMV; VFR; Peak systolic velocity; PSV; Peak velocity; PV; Neuromuscular electrical stimulation
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Intervention Model Description: All participants will be scanned, asked to use the NMES device for 30 minutes and scanned again.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Two ultrasound scans and activation of NMES device (Experimental): Participants will have their leg scanned using an ultrasound machine, before being asked to use the REVITIVE® device for 30 minutes. Their leg will then be scanned again.
  Interventions: Device: REVITIVE® device

INTERVENTIONS:
Device: REVITIVE® device — The REVITIVE® device applies neuromuscular electrical stimulation to the soles of the feet, causing the muscles of the leg to contract and relax, thus improving blood circulation through the legs.

SUMMARY:
The muscles of the leg require a regular supply of oxygen and nutrients. This is supplied by blood carried by a network of large blood vessels known as arteries. Gradually, these arteries can become narrowed or blocked by a build-up of fatty deposits. This process is known as atherosclerosis and leads to a condition called peripheral arterial disease. The restriction of blood flow caused by the blockage prevents exercising muscles getting enough oxygen and nutrients. In some people, this may lead to a painful ache in their legs when they walk, known as intermittent claudication. If the leg pain is severe, surgeons may decide to bypass this blockage using a vein taken from another part of the body, thereby improving blood flow to the foot.

Patients with a narrowing or blockage anywhere in the main artery that runs from the groin to the back of the knee may be treated with a particular type of bypass graft known as a femoral-popliteal bypass graft. However, this graft may collapse if not enough blood is flowing through it.

This study is looking to see whether a circulation booster machine, known as the REVITIVE® device, can improve the amount of blood flowing through femoral-popliteal bypass grafts. Patients with these grafts attending their usual clinic appointment in the Vascular Outpatients department at Charing Cross Hospital, London will be asked to have their leg scanned using an ultrasound machine to measure the amount of blood flowing through the graft. They will then use the REVITIVE® device for 30 minutes, before being re-scanned to see whether the device has improved blood flow. Improvements in blood flow may suggest a promising role for the device in keeping these grafts open, therefore helping them last longer and potentially reducing the leg pain associated with peripheral arterial disease.

DETAILED DESCRIPTION:
Within the vascular department at Charing Cross Hospital, there is an on-going NIHR-funded trial looking at the haemodynamics and clinical outcomes of patients with intermittent claudication. The aim of the study is to find out whether the neuromuscular electrical stimulation (NMES) device, REVITIVE®, can improve the time-averaged mean velocity (TAMV) and volume flow rate (VFR) through femoral-popliteal bypass grafts. Previous studies have shown that NMES can enhance arterial TAMV and VFR and have suggested the utility of NMES in the management of intermittent claudication, critical limb ischaemia and limb salvage. By enhancing arterial TAMV and VFR, NMES has been said to mimic the effect of exercise in the redistribution of arterial circulation. This is achieved through activation of the calf muscle pump, which empties the venous bed, thus increasing the pressure difference between the venous and arterial system. This creates a hyperaemic response in which there is faster arterial inflow against a lower venous back pressure. NMES could also enhance TAMV and VFR in femoral-popliteal bypass grafts which could, in turn, improve graft inflow and thus prolong patency.

If TAMV and VFR are enhanced, this may suggest that the REVITIVE® device could help prolong the patency of femoral-popliteal bypass grafts and be given to patients with these grafts to be used for 30 minutes daily as part of their management.

Methods

A Phillips (Guildford, UK) EPIQ 7 ultrasound machine and L12-5 transducer will be used to measure graft flow parameters using a pre-set optimised vascular protocol. A Phillips (Guildford, UK) EPIQ 7 ultrasound machine will be used as these are used frequently by Clinical Vascular Scientists in the Vascular Outpatients department to scan patients. An L12-5 transducer will be used as the proximal section of the femoral-popliteal graft will be scanned, which is a superficial structure and therefore a probe that is designed for imaging superficial structures should be used to obtain the best possible image resolution. Real-time gated Doppler superimposed on B-mode imaging will be used in the evaluation of flow and processed using automated waveform enveloping duplex software, as previously described.

First ultrasound scan: Patients will be called into a vascular ultrasound scanning room where a Clinical Vascular Scientist will ask the patient to rest for 10 minutes on an examination couch. A region of the femoral-popliteal bypass graft 3-5 cm from the saphenofemoral junction, or as proximal as possible depending on the patient's body habitus, will be identified and the position of the probe marked on the skin for consistency of repeat measurements. This method for maintaining consistency was chosen as it proved successful in similar studies. When obtaining measurements, the patient will be positioned semi-recumbent with the leg externally rotated at the hip to 35-40 degrees and flexed at the knee according to their comfort. Baseline measurements of TAMV and VFR (calculated using built-in software) will be taken and recorded via a 15-second electronic screenshot. All diameter measurements will be obtained by placing electronic callipers on the inner edge to inner edge of the graft to obtain the luminal diameter and to improve reliability of this measurement. Where indicated by reliability measurements (see below), a predetermined number of consecutive measurements of TAMV and VFR will be taken and an average calculated later. PV of the greatest waveform amplitude of each screenshot will be analysed at a later date using standard techniques.

Device activation: The REVITIVE® device will then be applied and activated for 30-minutes as per the instructions for use (IFU) of the device.

Second ultrasound scan: The Clinical Vascular Scientist will ask the patient to rest for another 10 minutes on the examination couch before performing a second ultrasound scan to obtain post-device TAMV and VFR measurements. The 10-minute equilibration periods were used in the study protocol as these were used in a similar study.

In order to determine the accuracy of measurements per subject (intrasubject reliability), 10 measurements each of TAMV, VFR and PSV will be performed the first five participants by the student (a trainee Clinical Vascular Scientist) on a marked region of the femoral-popliteal bypass graft. Data will be analysed to derive coefficient of variation, and Bland-Altman analysis will be performed (significance will be 0.05). To determine inter-user reliability, two different Clinical Vascular Scientists will each obtain 10 additional measurements of TAMV, VFR and PSV and Bland-Altman analysis performed again. Depending on the extent of variability of results, it may be decided to average at least three consecutive measurements of each variable. This will be applied to every patient in the study. These methods to assess reliability were chosen as these were used in similar studies.

Recruitment

The student, who is a member of the direct care team, will identify eligible patients and find their appointment information using Cerner, the health information system used by Imperial College Healthcare NHS Trust. Potential participants will be contacted in writing by the student before their next usual clinic appointment. The student will send out the patient information sheet along with the invitation letter, enabling the potential participant to read the about the study and discuss it with others. The student will also contact the potential participants by telephone to discuss the patient information sheet, explain the study further and allow the potential participant to ask questions if they wish.

At the patient's clinic appointment, the patient will have the opportunity to discuss the patient information sheet and the study further with a vascular physician. Female participants of child-bearing age will be asked whether or not they are pregnant - if they are, they will not be included in the study. If the patient is happy to take part in the study, they will be given a consent form to sign and the study intervention will be commenced and completed the same day. The patient will be given a copy of the consent form for their reference and reflection.

The study requires a sample size of 34 participants to achieve a power of 80% and a level of significance of 5% (two sided), for detecting an effect size of 0.5 between pairs [6]. An effect size of 0.5 was chosen as a previous study assessing VFR in arteries before and after NMES reported a 66% relative reduction with the test intervention (approximately 50%).

Consent

Obtaining valid consent enables healthcare professionals to act with beneficence towards their patients and to respect patient autonomy. The vascular physician will be seeking consent during the patient's clinic appointment. For consent to take part in the study to be valid, the patient must receive adequate information about the study, including risks and benefits, and have the capacity to decide for themselves. Through the patient information sheet and discussions with the patient, it will be ensured that the patient fully understands the purpose of the study and what it will involve for them. It will be ensured that any queries the patient may have are answered fully. The vascular physician will ask the patient if they have had the patient information sheet and study explained to them, and if their queries have been answered fully, before proceeding to take informed consent on the patient's decision. In keeping with the Mental Capacity Act 2005, all patients will be assumed to have capacity unless it is established otherwise.

When obtaining consent, the vascular physician will give the patient a personal anonymous identification number. This will be written on the patient's consent form and used throughout the study to anonymise the patient's personal and study data.

Risks and benefits

The REVITIVE® device is a commercially available, CE marked device which is intended to improve circulation. Therefore, it is expected that this study poses minimum safety risks provided that patients do not meet any of the exclusion criteria. Furthermore, extra precautions should be taken when using the device in certain individuals, for example those with a history of heart problems (the device may cause lethal rhythm disturbances to the heart in susceptible individuals) and with metallic implants. The long-term effects of chronic electrical stimulation are unknown; however the patients will be using the device for one 30-minute session only, which is well within the limit for the duration of use stated in the IFU (6 sessions of 30 minutes per day). Therefore, risks of muscle fatigue will be minimal.

The Philips EPIQ 7 ultrasound machine is used for the regular scanning of patients attending the Vascular Outpatients department at Charing Cross Hospital, London, therefore risks associated with use of the ultrasound machine are expected to be minimal. It will be ensured that the acoustic output intensity and mechanical index (MI) of the ultrasound machine is kept to within normal limits, thus minimising acoustic cavitation risk. The thermal index (TI) will also be kept to within normal limits, thus minimising tissue heating risk.

There could be benefits to the participants and other patients with femoral-popliteal grafts in the future because if the results show an improvement in blood flow through the femoral-popliteal grafts after use of the REVITIVE® device, the device may prolong graft patency if used in the longer-term. These patients could be offered the device to use daily. This study may inform future studies looking at the potential benefit of NMES on clinical outcomes in patients with PAD, including symptom relief and rehabilitation, which require some haemodynamic component in their analyses

Confidentiality

In line with the Caldicott Principles, person-identifiable information will only be used unless it is absolutely necessary. A document containing the participant's contact details such as their name, address and any medical information will be stored in a secure place, separate from any study data using the personal identification number. Contact details will be retained so that the participant can be contacted with a summary of the results once the study has ended, after which these documents will be disposed of in a confidential manner. Each participant will be assigned a personal anonymous identification number which will be written on the signed consent forms. Personal data will only be identified using the patient's anonymous identification number. Data obtained throughout the study (ultrasound measurements) will be stored on a password-protected electronic database. Only members of the study team will be able to access this and all data on the database will be identified using the patient's anonymous identification number only. Patients will not be identified from any study report or publication.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of peripheral arterial disease (PAD);
* Have undergone revascularisation surgery via a vein femoral-popliteal bypass graft;
* Are willing to participate and are able to provide written informed consent;
* Are aged over 18 years;
* Agree to attend at least one of their usual clinic appointments at the Vascular Outpatients department at Charing Cross Hospital, London before 13th April 2020 (project deadline for the student is Monday 11th May 2020);
* Have a body mass index (BMI) between 17 and 30 kg/m2.

Exclusion Criteria:

* Do not have a diagnosis of PAD;
* Have not had revascularisation surgery;
* Have had revascularisation surgery via an artificial femoral-popliteal bypass graft;
* Are fitted with an electronic implanted device;
* Are being treated for (or have symptoms of) a deep vein thrombosis (DVT);
* Are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Change in time-averaged mean velocity (TAMV). | 1 to 3 hours
  Change in TAMV in femoral-popliteal bypass grafts after use of the NMES device.
Change in peak systolic velocity (PSV). | 1 to 3 hours
  Change in PSV in femoral-popliteal bypass grafts after use of the NMES device.
Change in volume flow rate (VFR). | 1 to 3 hours
  Change in VFR in femoral-popliteal bypass grafts after use of the NMES device.

SECONDARY OUTCOMES:
Intra-subject reliability measurements of time-averaged mean velocity (TAMV). | 1 to 3 hours
  Intra-subject reliability measurements of TAMV will be made to determine the accuracy of measurements taken by the same operator.
Intra-subject reliability measurements of peak systolic velocity (PSV). | 1 to 3 hours
  Intra-subject reliability measurements of PSV will be made to determine the accuracy of measurements taken by the same operator.
Intra-subject reliability measurements of volume flow rate (VFR). | 1 to 3 hours
  Intra-subject reliability measurements of VFR will be made to determine the accuracy of measurements taken by the same operator.
Inter-user reliability measurements of time-averaged mean velocity (TAMV). | 1 to 3 hours
  Inter-user reliability measurements of TAMV will be made to determine the accuracy of measurements between operators.
Inter-user reliability measurements of peak systolic velocity (PSV). | 1 to 3 hours
  Inter-user reliability measurements of PSV will be made to determine the accuracy of measurements between operators.
Inter-user reliability measurements volume flow rate (VFR). | 1 to 3 hours
  Inter-user reliability measurements of VFR will be made to determine the accuracy of measurements between operators.

CONTACTS AND LOCATIONS:
Overall Officials: Alun H Davies, FHEA FACPh, Principal Investigator — Imperial College London
Locations (1):
- Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for the primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Access requests will be reviewed by the PI.

REFERENCES:
- [Background] Williams KJ, Moore HM, Davies AH. Haemodynamic changes with the use of neuromuscular electrical stimulation compared to intermittent pneumatic compression. Phlebology. 2015 Jun;30(5):365-72. doi: 10.1177/0268355514531255. Epub 2014 Apr 10. PMID 24722790
- [Background] Varatharajan L, Williams K, Moore H, Davies AH. The effect of footplate neuromuscular electrical stimulation on venous and arterial haemodynamics. Phlebology. 2015 Oct;30(9):648-50. doi: 10.1177/0268355514542682. Epub 2014 Jul 4. PMID 24997200
- [Background] Liu HI, Currier DP, Threlkeld AJ. Circulatory response of digital arteries associated with electrical stimulation of calf muscle in healthy subjects. Phys Ther. 1987 Mar;67(3):340-5. doi: 10.1093/ptj/67.3.340. PMID 2950528
- [Background] Ravikumar R, Williams KJ, Babber A, Lane TRA, Moore HM, Davies AH. Randomised Controlled Trial: Potential Benefit of a Footplate Neuromuscular Electrical Stimulation Device in Patients with Chronic Venous Disease. Eur J Vasc Endovasc Surg. 2017 Jan;53(1):114-121. doi: 10.1016/j.ejvs.2016.09.015. Epub 2016 Dec 2. PMID 27919609
- [Background] Delis KT, Knaggs AL, Sonecha TN, Zervas V, Jenkins MP, Wolfe JH. Lower limb venous haemodynamic impairment on dependency: quantification and implications for the "economy class" position. Thromb Haemost. 2004 May;91(5):941-50. doi: 10.1160/TH03-12-0754. PMID 15116255
- See also: Dhand, N.K. and Khatkar, M.S. (2014). Statulator: An online statistical calculator. Sample Size Calculator for Comparing Two Paired Means. — http://statulator.com/SampleSize/ss2PM.html